CLINICAL TRIAL: NCT05995288
Title: Homeopathic Treatment of Children Suffering From PFAPA: a Retrospective Case Series.
Brief Title: Homeopathic Treatment of Children Suffering From PFAPA
Acronym: HOMPFAPA
Status: Completed | Type: Observational
Sponsor: Michael Frass (Other)
Responsible Party: Sponsor-Investigator, Michael Frass, MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: 202308
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Periodic Fever Syndrome
Keywords: PFAPA; periodic fever; homeopathy; Naranjo criteria
MeSH Terms: conditions — Hereditary Autoinflammatory Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children suffering from PFAPA: Children suffering from periodic fever, with at least one of the following symptoms: aphthous stomatitis, pharyngitis, cervical adenitis
  Interventions: Drug: Homeopathic Globule

INTERVENTIONS:
Drug: Homeopathic Globule — Homeopathic globules were administered after careful anamnesis

SUMMARY:
Periodic fever, aphthous stomatitis, pharyngitis, cervical adenitis (PFAPA) syndrome is frequently diagnosed in young children. Fevers recurring at a nearly predictable rate every three to eight weeks are the signature symptom of PFAPA syndrome. PFAPA is an acquired autoinflammatory disorder, which recurs in association with at least one sign of aphthous stomatitis, pharyngitis, and cervical lymph node enlargement. The aim of this retrospective case report is to gain an impression of the course of disease during individualized homeopathic treatment in children suffering from PFAPA.

DETAILED DESCRIPTION:
In this retrospective study, the investigators collected the history and symptoms of 13 consecutive PFAPA patients. The investigators also described the individually chosen homeopathic medicinal products (HMPs) used, as well as the course of the disease. Clinical outcome of case reports was assessed using the "Modified Naranjo Criteria for Homeopathy-Causal Attribution Inventory". Eight points are taken as the threshold for the possible correlation between homeopathic therapy and improvement of symptoms or cure in chronic cases

ELIGIBILITY:
Inclusion Criteria:

Children suffering from fever with at least one of the symptooms of PFAPA besides fever

Exclusion Criteria:

Parents not willing to sign informed consent.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children were suffering from PFAPA for at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Periodic fever flares | 30 months
  Appearance of periodic fever flares

CONTACTS AND LOCATIONS:
Overall Officials: Peter Panhofer, MD, Study Director — Sigmund Freud Private University
Locations (1):
- Michael Frass, Vienna, Austria